CLINICAL TRIAL: NCT04644536
Title: Retrospective Collection of Safety and Performance Data
Status: Terminated | Type: Observational
Why Stopped: The study was terminated following a change in company management.
Sponsor: Bioceramed (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020.09
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Bone Defects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Granules in long bone & extremities: Filling of post-traumatic or surgically created bone defects
  Interventions: Device: Bone graft substitute
- Wedges in long bone & extremities: Osteotomies with fixation
  Interventions: Device: Bone graft substitute
- HA paste in long bone & extremities: Filling of post-traumatic or surgically created bone defects
  Interventions: Device: Bone graft substitute
- Granules in Spine: Spinal cage filling
  Interventions: Device: Bone graft substitute
- HA paste in Spine: Spinal cage filling
  Interventions: Device: Bone graft substitute

INTERVENTIONS:
Device: Bone graft substitute — Orthopaedic or Spine bony defects

SUMMARY:
This is a retrospective post market clinical follow-up study to compile real world clinical data on safety and efficacy of the synthetic bone graft substitutes in a commercial clinical setting in long bone and extremity defects and in spinal fusion procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with Bioceramed bone substitutes at the Center.
* Long bone & extremities: bone grafting after post-traumatic or surgically created bone defects.
* Spine: degenerative disc disease or trauma who require spinal fusion of 1 or more vertebral bodies.

Exclusion Criteria:

Serious infection within two months before surgery, active malignancy, cellulitis, osteomyelitis, diseases interfering with bone metabolism (primary hyperparathyroidism, severe renal or hepatic insufficiency, non-treated hyperthyroidism), other bone metabolic diseases (osteomalacia, Paget disease, osteogenesis imperfecta), bone metastasis, primary bone tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study patients will be extracted from current patient population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Bone healing, observable by x-ray/MRI | 6 months
  Primary endpoint will be successful radiographic bone repair.
Bone healing, observable by x-ray/MRI | 12 months
  Primary endpoint will be successful radiographic bone repair.

SECONDARY OUTCOMES:
Number and description of any adverse event during the follow-up | 6 - 12 months
  Record and description of any adverse event during the follow-up that reflects the safety of the bone graft substitute.

CONTACTS AND LOCATIONS:
Overall Officials: Nuno A Ribeiro, MD, Principal Investigator — Hospital Lusíadas Lisboa
Locations (1):
- Hospital Lusíadas Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No